CLINICAL TRIAL: NCT01108731
Title: The Effect of Milnacipran or Placebo on Ventricular Lactate Levels and Fibromyalgia Induced "Brain Fog."
Brief Title: The Effect of Milnacipran in Patients With Fibromyalgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIMC #212-09
Record Dates: First submitted 2010-03-30; First posted 2010-04-22 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2014-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients taking the drug Milnacipran (Active Comparator): Randomize patients signing informed consent and give 50% of them Milnacipran -- blinded to the investigators.
  Interventions: Drug: Milnacipran
- Patients taking the placebo (Placebo Comparator): Randomize patients signing informed consent and give 50% of them the placebo -- blinded to the investigators.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — Patients will take an increasing number of 12.5mg pills for the first 9 days during the "ramp up" period and then take one 50mg pill in the morning and one 50mg pill in the evening for the remaining 8 weeks of the study.
  Other Names: Savella
  Arms: Patients taking the drug Milnacipran
Drug: Placebo — Patients will take an increasing number of placebo pills for the first 9 days during the "ramp up" period and then take one pill in the morning and one in the evening for the remaining 8 weeks of the study.
  Arms: Patients taking the placebo

SUMMARY:
Use of the drug Milnacipran will reduce ventricular lactate levels and processing time for completing complex tasks relative to placebo.

DETAILED DESCRIPTION:
Patients with Fibromyalgia will show elevated ventricular lactate levels as measured via magnetic resonance spectroscopy (MRS). Patients treated with Milnacipran will show normalization of ventricular lactate levels compared to those treated with placebo, and will also show normalization of the increased latency to respond to complex reaction time probes compared to those treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects who fulfill the American College of Rheumatology's case definition for Fibromyalgia.
* 18 through 68 years of age

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Taking any other Serotonin Norepinephrine Reuptake Inhibitor (SNRI) or already taking milnacipran
* Patients who do not indicate their pain levels as less than substantial despite their best care
* History of any psychotic disorder or history of alcoholism or drug abuse within 10 years of intake as determined by psychiatric diagnostic interview
* Presence of current depression as determined by psychiatric diagnostic interview
* Presence of brain lesion on MRI anatomical study

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H Natelson, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Pain and Fatigue Study Center - Beth Israel Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natelson BH, Vu D, Mao X, Weiduschat N, Togo F, Lange G, Blate M, Kang G, Coplan JD, Shungu DC. Effect of Milnacipran Treatment on Ventricular Lactate in Fibromyalgia: A Randomized, Double-Blind, Placebo-Controlled Trial. J Pain. 2015 Nov;16(11):1211-9. doi: 10.1016/j.jpain.2015.08.004. Epub 2015 Aug 31. PMID 26335989
- See also: The Pain and Fatigue Study Center — http://www.painandfatigue.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We got informed consent from 37 patients but excluded 3 -- 2 for saving psychiatric diagnoses that were exclusionary and one for having a metal implant which was an exclusion for neuroimaging. Thus 34 patients were randomized for the trial.
Groups:
- Patients Taking the Drug Minalcipran: Milnacipran: Patients will take an increasing number of 12.5mg pills for the first 9 days during the "ramp up" period and then take one 50mg pill in the morning and one 50mg pill in the evening for the remaining 8 weeks of the study.
Period: Overall Study
Arm/Group | Patients Taking the Drug Minalcipran | Patients Taking the Placebo
Started | 17 | 17
Completed | 13 | 13
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 3 | 3

BASELINE CHARACTERISTICS:
Population: Had to report widespread pain and to have at least 11 of 18 tender points [rated on a 0 to 10 pain intensity scale at 2 or higher].
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Taking the Drug Minalcipran | Patients Taking the Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Age on intake, continuous
  years | 48 (4) | 47 (5) | 47 (4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Ventricular Lactate Levels in the Brain
Description: Ventricular lactate levels will be assessed before and at the end of the trial using a scanning method known as magnetic resonance spectroscopy (MRS), which is used to determine the presence and quantity of a number of chemicals in the brain.
Time Frame: Baseline and 2 months
Population: One drug treated and two placebo treated could not be analyzed due to excessive head motion
Measure: Mean (Standard Deviation); unit: international units (iu)
Arm/Group | Patients Taking the Drug Minalcipran | Patients Taking the Placebo
Number analyzed (Participants) | 12 | 11
international units (iu) | -0.87 (0.91) | 0.32 (1.58)
Statistical Analysis 1: Comparison: Patients Taking the Drug Minalcipran vs Patients Taking the Placebo; Test type: Superiority or Other; p < 0.05, General Linear Model (GLM)

2. Secondary Outcome: Change in Cognitive Function Assessed by the no Cue Condition of the Attention Network Test (ANT).
Description: The Attention Network Test (ANT) is a computerized test designed to evaluate the efficiency of the attention network. The ANT consists of a set of cued reaction time tasks to assess vigilance and efficiency to detect novel visual stimuli. The ANT also includes a set of flanker tasks during which a decision needs to be made about whether the orientation of a central stimulus is congruent or incongruent with a set of flanking arrows. Scores on the cued reaction time tasks (no cue, centre cue, double cue) reflect latency to respond measured in milliseconds (slower performance equals greater values). The score on the flanker task reflecting executive attention is derived by subtracting obtained latencies on the congruent flanker from the incongruent condition. Based on our prior work, we are hypothesizing that drug treated Ss will show improved performance on the no cue reaction time condition and on the derived executive attention variable compared to placebo treated.
Time Frame: Baseline and 2 months
Population: Data from 4 were excluded due to 2 having error rates greater than 50%, indicating that they did not understand the task and 2 having simple reaction times longer than those for the complex reaction times on the ANT, suggesting their need for additional practice trials on the simple motor reaction time task.
Measure: Mean (Standard Deviation); unit: latency to respond (msecs.)
Arm/Group | Patients Taking the Drug Minalcipran | Patients Taking the Placebo
Number analyzed (Participants) | 11 | 11
latency to respond (msecs.)
  No cue condition | -79.56 (80.45) | -35.00 (90.09)
  Executive attention | -68.73 (52.77) | -34.77 (52.77)
Statistical Analysis 1: Comparison: Patients Taking the Drug Minalcipran vs Patients Taking the Placebo; Test type: Superiority or Other; p < 0.05, General Linear Model (GLM)

3. Secondary Outcome: Change in Widespread Pain
Description: Pain was assessed using a visual analog scale (VAS) ranging from 0 (no pain) to 10 (worst pain ever). The baseline value recorded was widespread pain at the time of assessment and the 2 months follow value recorded was widespread pain over the week prior to assessment.
Time Frame: 2 months
Population: Data from all 26 participants were used for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Taking the Drug Minalcipran | Patients Taking the Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | -1.24 (1.57) | 0.66 (1.75)
Statistical Analysis 1: Comparison: Patients Taking the Drug Minalcipran vs Patients Taking the Placebo; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During the 2 month trial
Arm/Group | Patients Taking the Drug Minalcipran | Patients Taking the Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 2/17 | 1/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Taking the Drug Minalcipran (N=17) | Patients Taking the Placebo (N=17)
Gastric distress, nausea or vomiting (Gastrointestinal disorders) | 2 | 1 — A continuum of gastric distress, to nausea or frank vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes